CLINICAL TRIAL: NCT04421469
Title: A Single-arm, Open Multicenter Phase II Clinical Study of Triprilimab(JS001) and Chemotherapy Combined With Local Treatment for Multiple Metastatic NPC
Brief Title: Triprilimab(JS001) and Chemotherapy Combined With Local Treatment for Multiple Metastatic NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Zhejiang Cancer Hospital (Other); Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC005.1
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehensive treatment (Experimental): Patients with multiple metastatic NPC were given Triprilimab(JS001) and chemotherapy combined with local treatment.
  Interventions: Drug: Triprilimab(JS001)

INTERVENTIONS:
Drug: Triprilimab(JS001) — 1. JS001 240mg d1, gemcitabine(1g/m²),d1,8 + nedaplatin (80-100mg/m²),d2,q3w,6cycles.The curative effect was evaluated every 2 cycles.If the therapeutic evaluation was SD,the chemotherapy scheme was changed;
  2. Local treatment of active lesions(including radiotherapy and/or radiofrequency ablation);
  3. JS001 maintenance treatment.

SUMMARY:
This study is a randomized, phase II, prospective, multicenter clinical trial to evaluate the efficacy and tolerability of JS001 and chemotherapy combined with local treatment in patients with multiple metastatic nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with multiple metastases at first diagnosis or multiple metastases after treatment(multiple metastases was defined as more than 5 lesions and/or more than 2 metastasis organs); Histologically or cytologically confirmed multiple metastatic NPC.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at trial entry, and life expectancy ≥6months as judged by the Investigator;
3. The disease must be measurable with at least 1 unidimensional measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1;
4. Adequate organ function;
5. Take adequate contraceptive measures throughout the study, and contraception continues until 12 months after treatment;
6. Able and willing to provide signed informed consent form, and able to comply with all procedures.
7. The time from the last chemotherapy and/or radiotherapy to randomization must be ≥6 months.

Exclusion Criteria:

1. Patients with a hypersensitivity to any of the drugs used in our study;
2. With any active autoimmune disease or history of autoimmune disease;
3. Clinically significant cardiovascular and cerebrovascular diseases;
4. Have or are suffering from other malignant tumors within 5 years (except non-melanoma skin cancer or pre-invasive cervical cancer);
5. Active systemic infection;
6. Drug or alcohol abuse;
7. No or limited capacity for civil conduct;
8. The patient has a physical or mental disorder, and the researcher considers that the patient is unable to fully or fully understand the possible complications of this study;
9. History of immunodeficiency including seropositive for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or any active systemic viral infection requiring therapy；
10. Use cortisol or other systematic immunosuppressive medications within 4 weeks before the study treatment, and subject requiring hormone therapy during trials.
11. Pregnancy or breast feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival(PFS) | 2 year
  PFS was defined as the time from diagnosis of metastasis to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
ORR | 2 year
  Objective response rate
DCR | 2 year
  Disease contral rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China